CLINICAL TRIAL: NCT07332676
Title: Building Healthy Food Environment in Schools: Evaluating Co-created Interventions in Low Resource Settings. #BetterNutrition4Adolescent
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Institute for Implementation Science and Health (Unknown); Public Health Foundation of India (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 352614; 352614 (Other Grant/Funding Number: Research Council Norway)
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Overweight Adolescents; Underweight; Obese Adolescents
Keywords: nutrition; multicomponent nutrition intervention; co-creation; adolescent; low resource settings; Poor nutrition
MeSH Terms: conditions — Thinness; Malnutrition

STUDY DESIGN:
Intervention Model Description: We will utilise a hybrid type II approach to assess effectiveness and implementation using a parallel arm cluster RCT design with 12 months follow up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive co-created multicomponent school nutrition intervention and usual nutrition program (Experimental)
  Interventions: Other: Multicomponent school nutrition intervention
- Usual nutrition program (Active Comparator)
  Interventions: Other: Usual nutrition program

INTERVENTIONS:
Other: Multicomponent school nutrition intervention — The intervention will include innovative components that aims to change school food environment, nutrition education to promote healthy eating and community and parental involvement. This section will be completed after the intervention package is finalized during the co-creation phase.
  Arms: Receive co-created multicomponent school nutrition intervention and usual nutrition program
Other: Usual nutrition program — Usual nutrition program that is being implemented, no any additional active intervention
  Arms: Usual nutrition program

SUMMARY:
The goal of this clinical trial is to learn if a multicomponent nutrition program developed together with the students, parents, teachers and canteen operators will improve nutrition status of adolescents. It will also learn about the acceptability and feasibility of implementing the program in the school settings. The main questions it aims to answer are:

What is the effect of co-created multicomponent intervention promoting healthy food behavior and environment in schools on the proportion of normal weight adolescents? What proportion of the target adolescents and teachers does the intervention reach? What proportion of the schools are willing to implement the intervention? What was the level of fidelity of implementation of all components of the intervention and the barriers and facilitators to implementation? What is the cost for maintenance, and facilitators and barriers of sustainment? School going adolescents studying in grades 7 to 9 from 26 schools in India and 26 schools in Nepal will be enrolled in the trial and their height, weight, dietary behavior, mental well-being and physical activity will be measured at baseline and at 12 months follow up. After the baseline assessment the school community (students, school environment, parents, teachers, canteen operators) will receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents studying in grade 7 to 9 (aged 11-15 years) Exclusion criteria:

Exclusion Criteria:

* Adolescents with siblings enrolled in schools assigned to a different trial arm to avoid clustering, with underlying medical conditions and those who plan to change school within one year of enrollment (during follow up period) will be excluded.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2600 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of healthy weight adolescents and body mass index for age | At enrollment and at 12 months follow up
  Height and weight of the adolescents will be measured to calculate body mass index using age and sex specific charts and categorize them as Underweight: Less than the 5th percentile, Healthy weight: 5th percentile up to the 85th percentile , Overweight: 85th percentile to less than the 95th percentile, Obesity: 95th percentile or higher

SECONDARY OUTCOMES:
Total intake of fruits and vegetables, dairy products, meat and beans (protein), whole grains, sugar-sweetened beverages, fast food, and salty snacks | At enrollment and at 12 months follow up
  A 24 hour dietary recall will be taken (two times during week days and weekends)
Total metabolic equivalent per day (MET per day) | At enrollment and at 12 months follow up
  Use International Physical activity questionnaire for adolescent to measure specific types, frequency and duration across different domains.
Mental wellbeing | At enrollment and at 12 months follow up
  Measured using Warwick-Edinburgh Mental Well-Being Scale (WEMWBS)

CONTACTS AND LOCATIONS:
Overall Officials: Archana Shrestha, PhD, Principal Investigator — Institute for Implementation Science and Health; Monica Arora, PhD, Principal Investigator — Public Health Foundation India
Locations (2):
- Delhi, Delhi, India
- Budhanilakantha Municipality, Budhanilakantha, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No